CLINICAL TRIAL: NCT02202733
Title: A Caretaker Cooking Skills Intervention to Reduce Eating Out
Brief Title: Skill-based Cooking Intervention to Reduce Eating Out
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013-5379; Eating Out
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Obesity
Keywords: cooking skills; eating out; foods prepared away from home
MeSH Terms: conditions — Obesity | interventions — Cooking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cooking (Other): A skill-based cooking intervention for caretakers of an overweight/obese child aged 3-10 years.
  Interventions: Other: Cooking

INTERVENTIONS:
Other: Cooking — The aim is to test the feasibility of a skill-based cooking intervention to reduce the consumption of foods prepared away from home for the evening meal (e.g., pre-prepared frozen foods, restaurant foods, fast food, take-out), energy intake from evening meals, and parent/child weight status.

SUMMARY:
The primary goal of the study is to use an iterative process to develop and refine a skill-based cooking intervention to decrease the consumption of energy from foods prepared away from home for evening meals, decrease energy intake, and promote a healthy weight in parents and children aged 3-10 years.

DETAILED DESCRIPTION:
Phase I. Conduct 2-4 focus groups with 6-10 caretaker, who report eating foods prepared away from home ≥3 times per week, per group to gain insight into current eating behaviors of foods prepared away from home, current perceptions about a home prepared evening meal, and barriers to preparing evening meals at home. Information gathered during Phase I will be used to inform intervention development in Phase II.

Phase II. Develop, refine, and manualize a skill-based cooking intervention for overweight/obese caretakers of a child aged 3-10 years. The aim of Phase II is to test the feasibility of a skill-based cooking intervention to reduce the consumption of foods prepared away from home for the evening meal (e.g., pre-prepared frozen foods, restaurant foods, fast food, take-out), energy intake from evening meals, and promote a healthy weight in parents and children. Information collected during Phase I will inform the development of the skill-based cooking intervention. Once developed, the intervention will be refined with 6 primary caretakers of a child, who meet criteria for being overweight/obese during a testing phase. Conducting the intervention with at least six families will provide the opportunity for further refinement of intervention procedures. The results will be important to demonstrate feasibility for a future pilot randomized controlled trial that will test the impact of a skill-based cooking intervention compared to a standard cooking demonstration where recipes are simply provided to families.

ELIGIBILITY:
Inclusion Criteria (Phase I):

* be ≥18 years of age
* have a child between the ages of 3 and 10 years-old
* report being the primary caretaker and have the primary feeding responsibility of the child for dinner/supper
* able to read, speak, and understand English
* have transportation to the Medical Center
* report their family including the child eats pre-prepared frozen food, restaurant food, fast food, or take-out for dinner ≥3 times per week
* has a working telephone number
* is able to attend the scheduled date and time of a focus group.

Inclusion Criteria (Phase II):

* caretaker is ≥18 years of age
* caretaker is overweight or obese (BMI≥25)
* has a child between the ages of 3 and 10 years-old
* report being the primary caretaker and have the primary feeding responsibility of the child for dinner/supper
* caretaker is able to read, speak, and understand English
* has transportation to the medical center and the instructional kitchen
* does not plan to move out of the area before June 2015
* reports their family including the child eats convenience food, restaurant food, fast food, or take-out for dinner ≥3 times per week
* reports access to a kitchen
* able to attend the scheduled date and time of the sessions.

Exclusion Criteria (Phase II):

* the caretaker or child is currently participating in a weight loss program and/or taking weight loss medication
* have a medical condition known to promote growth (e.g., Prader-Willi syndrome, Cushing's syndrome) or had gastric bypass surgery.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Dietary Intake (Phase II only) | 0 and 10 weeks
  Caregivers will be asked to complete a 7-day dietary record of what they and their child eat at the evening meal. For each evening meal, the caretaker will be asked to describe the meal type (fast food, restaurant, pre-prepared frozen meal, or home prepared); the specific foods and drinks consumed, and the amount consumed by the child. Data from dietary records will be input into Nutrition Data System for Research (NDSR) software and analyzed for energy intake, percent energy from fat, and food groups (fruits, vegetables, grains, proteins, dairy) from the evening meal. Foods prepared away from home will be classified based on caretaker indication of fast food, restaurant, pre-prepared frozen meal, or home prepared on the dietary record.

SECONDARY OUTCOMES:
Caretaker Attitudes and Confidence | 0 and 10 weeks
  Caretakers will report ease of providing foods prepared away from home (i.e., pre-prepared frozen meals, restaurant food, fast food, take-out) for an evening meal, ease of providing a home prepared evening meal, and their confidence with meal preparation using a 100-mm visual analog scale (VAS). Further caretakers will rate their ability, enjoyment of cooking and desire to cook on a 100-mm VAS.
Food Costs | 0 and 10 weeks
  Caretakers will be provided with four visual images with each image showing one adult evening meal and two child evening meals. Caretaker will record the total cost of the meals shown in each image.
Portions | 0 and 10 weeks
  Caretakers will be provided with visual images of foods in different portion amounts and asked to identify which image best represents the amount their child would be served for dinner. Caretakers will also identify the images that best represent the amount they would serve themselves for dinner.
Dinner Choices | 0 and 10 weeks
  Caretakers will complete a 10-question, open-ended questionnaire that solicits information related to choices of foods prepared away from home and foods prepared at home.
Anthropometrics | 0 adn 10 weeks
  Height and weight will be measured using standard procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States